CLINICAL TRIAL: NCT03016234
Title: Intraocular Pressure Changes During Laparoscopic Colorectal Surgery: Propofol Versus Desflurane Anesthesia
Brief Title: IOP Changes With Different Anesthetic Agents During Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Seo, Kwon Hui, Clinical Assistant Professor, Department of anesthesia and pain medicine, Saint Vincent's Hospital, Korea, Saint Vincent's Hospital, Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VC16OISI0143
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Intraocular Pressure
Keywords: intraocular pressure; trendelenburg position; pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum | interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane (Active Comparator): inhalation anesthesia administration for maintenance of anesthesia
  Interventions: Drug: Desflurane
- Propofol (Active Comparator): intravenous anesthesia administration for maintenance of anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desflurane — On arrival in the operating room, initial intraocular pressure is measured after administration of alcaine 0.5% eye drop and routine monitoring and bispectral index(BIS) are applied. Anesthesia is induced with pentothal sodium inj (thiopental sodium 0.53g) 5-6mg/kg and esmeron inj (rocuronium bromide 50mg/5ml) 1mg/kg. Then endotracheal intubation is performed, anesthesia is maintained with 50% oxygen-air-4~7% desflurane inhalation and intravenous remifentanil continous infusion (effect site concentration 3-6ng/mL) during operation. Desflurane concentration is titrated to maintain BIS values within a target range 40-60 during operation. Mean arterial blood pressure, peak airway pressure, end tidal carbon dioxide, and IOP on both eyes are measured at defined intervals.
  Other Names: Suprane soln. 240ml/Bottle
  Arms: Desflurane
Drug: Propofol — On arrival in the operating room, initial intraocular pressure is measured after administration of alcaine 0.5% eye drop and routine monitoring and bispectral index(BIS) are applied. Anesthesia is induced with fresofol MCT 1% inj (1% propofol) 1.5-2.5mg/kg and esmeron inj (rocuronium bromide 50mg/5ml) 1mg/kg. Then endotracheal intubation is performed, anesthesia is maintained with intravenous fresofol MCT 2% inj (2% propofol, effect site concentration 2.5-5μg/mL) and remifentanil (effect site concentration 3-6ng/mL) continous infusion. Effect site concentration of propofol is titrated to maintain BIS values within a target range 40-60 during operation. Mean arterial blood pressure, peak airway pressure, end tidal carbon dioxide, and IOP on both eyes are measured at defined intervals.
  Other Names: Fresofol medium-chain triglyceride (MCT) 2% inj. 50mL
  Arms: Propofol

SUMMARY:
This study is aimed to evaluate how intraocular pressure (IOP) is changed depending on surgical position (Trendelenburg versus reverse Trendelenburg) in the same patient and to compare the effects of different anesthetics on IOP (desflurane versus propofol) in patients undergoing laparoscopic colorectal surgery. The study design is a double-blind randomized controlled trial. The patients were randomly assigned to desflurane or propofol administrated groups and all patient are administered intravenous remifentanil continuously as adjuvant analgesics during anesthesia. For this study 50 to 80-year-old patients undergoing laparoscopic colorectal surgery without eye disease were enrolled. Mean arterial blood pressure, peak airway pressure, end tidal carbon dioxide, and IOP (using a Tono-pen® Avia tonometer) on both eyes were measured at defined intervals during the procedure.

DETAILED DESCRIPTION:
Perioperative visual loss is a rare but devastating complication associated with certain type of operative procedures. Laparoscopic or robotic surgeries for colorectal cancer, prostate cancer and diseases of the female genital organs in the pelvic cavity are performed in a steep Trendelenburg position and pneumoperitoneum, which increases the intraocular pressure (IOP) by 13-26 mmHg compared with the preoperative IOP value. High intraocular pressure is believed to correlate with decreased perfusion to the optic nerve, and thus could lead to ischemic optic neuropathy. The objective of the study is to test which anesthetic agent (desflurane or propofol) can attenuate the changes in IOP during laparoscopic colorectal surgery and identify correlated parameters. Fifty patients (30-80 years; American Society of Anesthesiologists' physical status 1-2) scheduled for laparoscopic colorectal surgery will be enrolled and allocated randomly into two groups (group D and group P). After measurement of initial IOP with topical opthalmic anesthetics, general anesthesia will be induced with pentothal sodium 5-6mg/kg (group D) or propofol (group P) 2-2.5mg/kg. After administration of muscle relaxant and intubation, intraocular pressure will be measured and anesthesia will be maintained with desflurane (group D) or propofol (group P) and all patients will be administered intravenous remifentanil concurrently during anesthesia. During anesthesia, IOP will be measured at different patient positions. At the time of each IOP measurements, the following data set will be collected: mean arterial pressure (MAP), End tidal carbon dioxide (EtCO2), peak inspiratory pressure (PIP).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopic colorectal surgery American society of anesthesiologist physical status class I or II

Exclusion Criteria:

* opthalmic disease or previously undergone opthalmic surgery, uncontrolled hypertension, arrythmia, psychiatric disorder, uncontrolled obstructive lung disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
changes in intraocular pressure (IOP) in different positions during laparoscopic colorectal surgery under desflurane or propofol anesthesia. | before anesthesia induction, immediately after intubation, after pneumoperitoneum, 30 minutes after head down and right tilt position, 10 minutes after head up and right tilt, 30 minutes after head down and right tilt and 5 minutes before extubation
  T1 (baseline: initial IOP before anesthesia induction), T2 (immediately after endotracheal intubation), T3(after pneumoperitoneum in supine position), T4 (30 minutes after position change to head down and right tilt), T5 (10 minutes after position change to head up and right tilt), T6 (30 minutes after position change to head down and right tilt) and T7 (5 minutes before endotracheal extubation)

SECONDARY OUTCOMES:
changes in mean arterial pressure (MAP) in different positions during laparoscopic colorectal surgery under desflurane or propofol anesthesia. | before anesthesia induction, immediately after intubation, after pneumoperitoneum, 30 minutes after head down and right tilt position, 10 minutes after head up and right tilt, 30 minutes after head down and right tilt and 5 minutes before extubation
  T1 (baseline: initial MAP before anesthesia induction), T2 (immediately after endotracheal intubation), T3(after pneumoperitoneum in supine position), T4 (30 minutes after position change to head down and right tilt), T5 (10 minutes after position change to head up and right tilt), T6 (30 minutes after position change to head down and right tilt) and T7 (5 minutes before endotracheal extubation)
changes in end tidal carbon dioxide in different positions during laparoscopic colorectal surgery under desflurane or propofol anesthesia. | immediately after intubation, after pneumoperitoneum, 30 minutes after head down and right tilt position, 10 minutes after head up and right tilt, 30 minutes after head down and right tilt and 5 minutes before extubation
  T2 (immediately after endotracheal intubation), T3(after pneumoperitoneum in supine position), T4 (30 mins after position change to head down and right tilt), T5 (10 mins after position change to head up and right tilt), T6 (30 mins after position change to head down and right tilt) and T7 (5 minutes before endotracheal extubation)
changes in peak airway pressure in different positions during laparoscopic colorectal surgery under desflurane or propofol anesthesia. | immediately after intubation, after pneumoperitoneum, 30 minutes after head down and right tilt position, 10 minutes after head up and right tilt, 30 minutes after head down and right tilt and 5 minutes before extubation
  T2 (immediately after endotracheal intubation), T3(after pneumoperitoneum in supine position), T4 (30 mins after position change to head down and right tilt), T5 (10 mins after position change to head up and right tilt), T6 (30 mins after position change to head down and right tilt) and T7 (5 minutes before endotracheal extubation)

CONTACTS AND LOCATIONS:
Overall Officials: Kwon hui Seo, MD, Principal Investigator — Saint Vincent's Hospital, Korea
Locations (1):
- Saint Vincent's Hospital, Korea, Suwon, Gyonggido, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Joo J, Koh H, Lee K, Lee J. Effects of Systemic Administration of Dexmedetomidine on Intraocular Pressure and Ocular Perfusion Pressure during Laparoscopic Surgery in a Steep Trendelenburg Position: Prospective, Randomized, Double-Blinded Study. J Korean Med Sci. 2016 Jun;31(6):989-96. doi: 10.3346/jkms.2016.31.6.989. Epub 2016 Apr 6. PMID 27247511